CLINICAL TRIAL: NCT02970487
Title: Refractive Outcome and Optimization of IOL-Constants After Implantation of the Precisight® Intraocular Lens.
Brief Title: Precisight® Intraocular Lens Implantation for Cataract Treatment
Acronym: PEACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InfiniteVision Optics (Industry)
Collaborators: Targomed (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0023
Record Dates: First submitted 2016-11-10; First posted 2016-11-22 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Cataract Senile
Keywords: cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- investigational device (Experimental): Subjects implanted with the Precisight intraocular lens.
  Interventions: Device: Intraocular implant of the Precisight

INTERVENTIONS:
Device: Intraocular implant of the Precisight — Precisight ismplanted in place of the natural cloudy lens, inside the capsular bag.

SUMMARY:
The purpose of this study is to determine the refractive outcomes and optimize the clinical features of a new intraocular lens intended to treat the senile cataract.

DETAILED DESCRIPTION:
InfiniteVision Optics has developed a new IOL system, the Precisight IOL. This IOL consists of a combination of two lenses: a base lens which is placed permanently into the capsular bag, and a front lens which sits on top of the base lens outside the capsular bag. The major advantage of this system is the adjustability of the primary IOL implantation which is done by front lens exchange. In case of either postoperative refractive adjustments or patient dissatisfaction with the visual performance, the front lens can be easily exchange by a less invasive surgery, avoiding a total IOL explantation. The implantation of the Precisight IOL is similar to the implantation of a traditional intraocular lens with no expected additional risk.

For all new IOLs, the IOL-constants are determined and provided by the manufacturer. They are calculated on the basis of eye models and clinical testing. In this study the biometric data of each patient's eye will be documented together with the implanted lens power and the postoperative stable refraction for calculation of the optimized IOL-constants.

In the present study, 125 subjects will be enrolled. Patients with a deviation from target refraction of more than 0.5 D spherical equivalent at the 2-3 month follow-up visit will undergo a secondary intervention for exchange of the front lens. These patients will be followed up for 1 year after front lens exchange.

Subjects will be screened during a pre-operative visit. Before the surgery visit, the subjected must have signed the Informed Consent Form.

After the surgery, patients will be followed up for one year. The visits will be scheduled at 1 day, 7-14 days, 2-3 months and 5-7 months and 1 year after surgery. Patients who underwent a surgery to exchange the front lens will be also followed up 1 day, 7-14 days, 2-3 months and 5-7 months and 1 year after the exchange surgery.

Investigator site staff will document the data in electronic Case Report Forms (eCRF). The data will be pseudonymized, i.e. only the year of birth and a code will be entered in the eCRF. Adverse events will be recorded in an eCRFs. Unexpected and serious adverse events are to be reported to the manufacturer.

Data cleaning will be done one month after last patient out and study report finished three months after last patient out. Subjects must be withdrawn from the study (i) at their own request, (ii) in case of intraoperative complication impacting the safety of the patient or (iii) in case of any postoperative complication if the continuation of the study has an impact on the safety of the patient. The study may terminate before completion if a high relative number of individual subject withdrawals due to the patient's requests and/or clinically relevant complications are observed. The IRB will be informed in due course accordingly.

The findings of this study will be published by the investigators in a scientific journal and presented at scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Age-related bilateral cataract or one pseudophakic eye
* Visual acuity potential of the study eye of at least 0.63 (decimal)
* Expected postoperative astigmatism of ≤0.75 D in the study eye
* IOL power within available diopters
* Written informed patient consent regarding participation in the study and data protection

Exclusion Criteria:

* Visually significant corneal scars
* Ocular disorders - other than cataract - that could potentially cause future acuity losses to a level of 0.5 (decimal) or worse in the study eye
* Relevant concomitant ophthalmic diseases (such as pseudoexfoliation, angleclosure glaucoma, traumatic cataract and other co-morbidity that could affect capsular bag stability (e.g. Marfan syndrome)
* Participation of patient in other clinical trials (former participation is not an exclusion criterion)
* Any cataract condition that makes the assessment of retina status difficult
* Anyone with unstable systemic conditions or untreated systemic medical problems including but not limited to the following: Untreated diabetes, Cardiovascular untreated disease, Pulmonary untreated disease, Any untreated infection, Neuro-ophthalmologic diseases, Any allergy to the medications used during surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-06; Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change of the subjective refraction | 2 to 3 months, 5 to 7 months and 1 year after the investigational device implantation
  The evolution of subjective refraction will be assessed after Precisight implantation.

SECONDARY OUTCOMES:
Best-corrected distance visual acuity | 1 day, 7 to 14 days, 2 to 3 months, 5 to 7 months and 1 year after the investigational device implantation
Introcular lens (IOL) decentration and tilt | day of surgery, 2 to 3 months, 5 to 7 months and 1 year after the investigational device implantation
Anterior chamber depth | pre-operative, 2 to 3 months, 5 to 7 months and 1 year after the investigational device implantation
Adverse events | All follow up period (1 year)
Assessment of investigator regarding handling and achievement of target refraction | Six months after investigational device implantation
  The investigator shall answer a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Uy, MD, Principal Investigator — Peregrine Eye and Laser Institute
Locations (1):
- Peregrine Eye and Laser Institue, Makati, Philippines

IPD SHARING:
Plan to Share IPD: No